CLINICAL TRIAL: NCT01662219
Title: Effect of Superficial Cervical Plexus Block on the Postoperative Quality of Recovery After Anterior Cervical Discectomy and Fusion
Brief Title: Effect of Superficial Cervical Plexus Block on the Postoperative Quality of Recovery
Acronym: QoR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Lashmi Venkatraghavan, Dr. Lashmikumar Venkatraghavan, Asst. Professor,Dept. of Anesthesia, TWH, UHN,Toronto,ON., University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-0210-A
Record Dates: First submitted 2012-07-24; First posted 2012-08-10 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Cervical Disc Prolapse
Keywords: superficial cervical plexus block; quality of recovery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- superficial cervical plexus block (Experimental): superficial cervical plexus block for experimental group
  Interventions: Other: Superficial cervical plexus block for experimental group
- No Block (No Intervention): no superficial cervical plexus block for the no intervention group

INTERVENTIONS:
Other: Superficial cervical plexus block for experimental group — 15 ml of 0.25% Bupivacaine will be given for superficial cervical plexus block
  Arms: superficial cervical plexus block

SUMMARY:
Pain and discomfort after anterior cervical spine surgery is difficult to quantify and quoted as moderate in severity, often needing oral opioid analgesics. In addition, these patients are more prone for postoperative respiratory complication due to airway edema secondary to surgical retraction or wound hematoma. Opioid analgesics provide good pain control but postoperative nausea and vomiting and respiratory depression are undesirable in these patients who are at risk for postoperative wound hematoma and airway edema The use of multimodal analgesia is rapidly becoming the 'standard of care' for preventing pain after ambulatory procedures at most surgery centers throughout the world . The purpose of this study is to determine whether superficial cervical plexus block will improve the postoperative quality of recovery as measured by Quality of Recovery 40 questionnaire (QoR-40) in patients undergoing elective anterior cervical discectomy and fusion.

DETAILED DESCRIPTION:
Anterior cervical discectomy and fusion is increasingly being done as a day surgery or short stay surgery. Postoperative pain is the leading cause of unplanned hospital admissions following day surgery, a major source of dissatisfaction and often impairs the quality of recovery. Opioid analgesics alone are not always effective and may also worsen the postoperative nausea and vomiting and in turn the postoperative recovery. This study is designed to find out if an injection of freezing on the side of neck around the nerves (superficial cervical plexus block) improves the quality of recovery from anesthesia and surgery by reducing the pain, analgesic consumption after anterior cervical spine surgery.

Primary Outcome Measure The primary outcome measure is the global QoR-40 aggregate score at 24 hours after surgery.

Secondary Outcome Measures

* Postoperative pain scores (first 24 hours)
* Total analgesic consumption (first 24 hours)
* Time for first opioid administration
* Postop Nausea and vomiting (first 24 hours)
* Post operative sedation (first 24 hours)

ELIGIBILITY:
Inclusion Criteria:

* all adult patients
* aged 18-80 years
* with ASA class I - III
* undergoing anterior cervical disc surgery in supine position

Exclusion Criteria:

1. In patients who are allergic to local anesthetics
2. ASA- IV patients
3. Lack of informed consent
4. Pregnant patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the global QoR-40 aggregate score after ACDF surgery. | 24 hours

SECONDARY OUTCOMES:
post operative pain score assessment | 24 hours
Post operative analgesic consumption | 24 hours
time for the first dose of opioid consumption | 24 hrs
post operative nausea and vomiting | 24 hrs
post operative sedation score | 24 hrs

CONTACTS AND LOCATIONS:
Overall Officials: lashmikumar venkatraghavan, MD, Principal Investigator — TWH,UHN,Toronto Canada
Locations (1):
- Toronto Western Hospital,UHN., Toronto, Ontario, Canada

REFERENCES:
- [Derived] Mariappan R, Mehta J, Massicotte E, Nagappa M, Manninen P, Venkatraghavan L. Effect of superficial cervical plexus block on postoperative quality of recovery after anterior cervical discectomy and fusion: a randomized controlled trial. Can J Anaesth. 2015 Aug;62(8):883-90. doi: 10.1007/s12630-015-0382-3. Epub 2015 Apr 14. PMID 25869024